CLINICAL TRIAL: NCT01941342
Title: Evaluation of Preoperative Biliary Drainage on Outcome of Pancreatoduodenectomy: A Multicenter Randomized Controlled Study
Brief Title: Evaluation of Preoperative Biliary Drainage Before Pancreatoduodenectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Huai-zhi Wang, Doctor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NDR-2014-02
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer; Periampullary Carcinoma
Keywords: Obstructive Jaundice; Preoperative Biliary Drainage; Pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Jaundice, Obstructive | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pancreatoduodenectomy (Active Comparator): Instant pancreatoduodenectomy within one week after diagnosis including: Evaluate the resectability; Remove pancreas head, gastric pyloric antrum, duodenum, distal common bile duct and regional lymph nodes; Reconstruct digestive tract.
  Interventions: Procedure: Pancreatoduodenectomy
- ENBD and Pancreatoduodenectomy (Experimental): Consistent ENBD (Endoscopic Nasobiliary Drainage) for 3 weeks or drainage until bilirubin level decreases to 200μmol per liter or below then perform pancreatoduodenectomy including:
  Evaluate the resectability; Remove pancreas head, gastric pyloric antrum, duodenum, distal common bile duct and regional lymph nodes; Reconstruct digestive tract.
  Interventions: Procedure: ENBD and Pancreatoduodenectomy
- EBD and Pancreatoduodenectomy (Experimental): Consistent EBD (Endoscopic Biliary Drainage) for 3 weeks or drainage until bilirubin level decreases to 200μmol per liter or below then perform pancreatoduodenectomy including:
  Evaluate the resectability; Remove pancreas head, gastric pyloric antrum, duodenum, distal common bile duct and regional lymph nodes; Reconstruct digestive tract.
  Interventions: Procedure: EBD and Pancreatoduodenectomy
- PTCD and Pancreatoduodenectomy (Experimental): Consistent PTCD (Percutaneous Transhepatic Cholangial Drainage) for 3 weeks or drainage until bilirubin level decreases to 200μmol per liter or below then perform pancreatoduodenectomy including:
  Evaluate the resectability; Remove pancreas head, gastric pyloric antrum, duodenum, distal common bile duct and regional lymph nodes; Reconstruct digestive tract.
  Interventions: Procedure: PTCD and Pancreatoduodenectomy

INTERVENTIONS:
Procedure: Pancreatoduodenectomy
  Arms: Pancreatoduodenectomy
Procedure: ENBD and Pancreatoduodenectomy
  Arms: ENBD and Pancreatoduodenectomy
Procedure: EBD and Pancreatoduodenectomy
  Arms: EBD and Pancreatoduodenectomy
Procedure: PTCD and Pancreatoduodenectomy
  Arms: PTCD and Pancreatoduodenectomy

SUMMARY:
The purpose of this study is to evaluate the efficacy of preoperative biliary drainage (PBD) which is performed prior to pancreatoduodenectomy candidates with obstructive jaundice by observing the prevalence of drainage and surgery related complications, hospital stay, medical cost and life quality compared to surgery alone. It is anticipated that PBD can reduce the prevalence of complications and improve the outcome of pancreatoduodenectomy.

DETAILED DESCRIPTION:
Obstructive jaundice is a common symptom in patients with pancreatic head cancer or peri-ampullary cancer. It is regarded that proper surgical resection is the only possible way of radical cure for those patients without evidence of metastasis. Since high preoperative bilirubin level is suggested to be a risk factor for pancreatoduodenectomy, preoperative biliary drainage has been applied to clinical practice to improve the outcome of surgery. However, results from previous studies have inconsistent results showing that PBD may have adverse effect on patients by elevating the prevalence of complications. Since PBD is widely performed worldwide, its value needs to be clarified. Thus the present study is designed to systematically evaluate the value of PBD via recruiting participants who may most likely benefit from PBD. It is anticipated that results from this study can present an instructive conclusion on whether PBD should be performed prior to pancreatoduodenectomy as well as reveal the preferable type of PBD.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* CT (Computed Tomography), CTA (Computed Tomographic Angiography), MRI (Magnetic Resonance Imaging) or ultrasonic test suggested pancreatic head carcinoma or periampullary carcinoma with obstructive jaundice
* First routine test of serum bilirubin above 250μmol per liter

Exclusion Criteria:

* Distant metastasis in liver, lung or other sites
* Invasion of local blood vessels (e.g. aorta, portal vein, postcava)
* Poor physical condition, unable to tolerate anesthesia and surgery (e.g. severe cardio-pulmonary diseases, blood coagulation disorders)
* With cholangitis, active hepatitis or other diseases which should be excluded from study according to the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Infectious Complications | up to 12 months

SECONDARY OUTCOMES:
Incidence of Hemorrhagic Complications | up to 6 months
Liver Function Evaluation | up to 6 months
Incidence of Bile Leakage | up to 6 months
Incidence of Pancreatic Leakage | up to 6 months
Life Quality Score | up to 12 months
Digestive Function Recovery | up to 6 months

OTHER OUTCOMES:
Incidence of Incision Complications | up to 3 months
Incidence of Pulmonary Infections | up to 6 months
Incidence of Pleural Effusion | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Huai-zhi Wang, M.D., Ph.D., Principal Investigator — Southwest Hospital, China
Locations (1):
- Institution of Hepatobiliary Surgery, Southwest Hospital, Chongqing, Chongqing Municipality, China